CLINICAL TRIAL: NCT03217240
Title: Integrated Computational modelIing of Right Heart Mechanics and Blood Flow Dynamics in Congenital Heart Disease ("INITIATE")
Brief Title: Integrated Computational modelIng of Right Heart Mechanics and Blood Flow Dynamics in Congenital Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: NHeartCentreS
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Congenital Heart Disease; Pulmonary Hypertension
MeSH Terms: conditions — Heart Defects, Congenital; Hypertension, Pulmonary | interventions — Exercise Test; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples will be obtained before CMR. The sample will be stored at -80 degree until assay. Investigators will perform various tests related to participants heart function
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Congenital Heart Disease: Tetralogy of Fallot Repair/Pulmonary Hypertension Cardiac Magnetic Resonance - MRI Cardiopulmonary Exercise Test Blood Sampling for all participants
  Interventions: Procedure: Cardiac Magnetic Resonance - MRI; Other: Cardiopulmonary Exercise Test; Other: Blood Sampling for all participants
- Healthy Volunteer: Cardiac Magnetic Resonance - MRI Cardiopulmonary Exercise Test Blood Sampling for all participants
  Interventions: Procedure: Cardiac Magnetic Resonance - MRI; Other: Cardiopulmonary Exercise Test; Other: Blood Sampling for all participants

INTERVENTIONS:
Procedure: Cardiac Magnetic Resonance - MRI — All participants will have to undergo CMR which uses interaction of the magnetic properties of body tissues with strong magnetic fields to create images. Participants will be asked to lie on a narrow bed placed inside of a large magnet for about 1 hour. Several sets of images are needed. Participants are required to stay very still and follow the instruction of the MRI technologist who operates the machine from a room next door.
Other: Cardiopulmonary Exercise Test — Participants will be asked to undergo a cardiopulmonary exercise test (CPET). Participants will need to wear a mask. Several electrodes will be placed on the chest to record heart activity during exercise. Participants will need to pedal for at least 8-12 minutes. Pedalling will be instructed to report any symptoms such as chest discomfort, shortness of breath, leg fatigue or dizziness. A small probe will be placed on participant's finger during the test to measure the oxygen content in the blood. Immediately after exercising, participants will rest for 5-10 minutes while the blood pressure and electrocardiogram are monitored. The results will be read by a cardiologist.
Other: Blood Sampling for all participants — Serum samples will be obtained before CMR. The sample will be stored at -80 degree until assay. Investigators will perform various tests related to participants heart function

SUMMARY:
Advances in paediatric cardiology and cardiac surgery have enabled the survival of most patients born with congenital heart disease (CHD) into adulthood. Many CHD patients have undergone palliative or reparative surgery earlier in life. As patients survive into adulthood, they may need intervention or surgery for residual haemodynamic lesions. This is because they are at risk of arrhythmias secondary to structure heart disease and are susceptible to acquired heart disease. In these patients, pre-operative and post-operative evaluation of right ventricular (RV) structure (shape and volume) and function is an essential component of clinical management.

Advances have been made in cardiac imaging so that accurate assessment of the right heart chamber in terms of its structure, function and physiology is possible. However, this technology has as yet never been applied in an effort to comprehensively assess RV structure, function and physiology. Cardiac Magnetic Resonance (CMR) will be used in this comprehensive assessment of structure and function. Thus, this research will allow development of a comprehensive integrated biomedical engineering (BME) R&D platform for in-depth study and clinical diagnosis of the RV structure-function relationship and physiology and its association with biomarker, and exercise capacity in CHD.

DETAILED DESCRIPTION:
The incidence of Congenital Heart Disease (CHD) in live new-borns is estimated to vary from 4.1/1000 to 12.3/1000. The improvement in survival of CHD patients has led to burgeoning numbers of grown-up CHD.The majority of these CHD patients face a lifetime of problems including RV dilation, ventricular arrhythmias, and sudden cardiac death.Considering inflation to visit costs and added image technology for diagnosis, the cost of each patient is expected to increase .In contrast to adult patients with acquired heart disease, abnormalities of the RV are ubiquitous in children and adults with CHD.

Currently, clinical evaluation includes ECG and pulse oximetry alongside clinical examination. Investigation of RV anatomy and physiology is evolving from a reliance on invasive studies (right heart catheterization or RHC) to non-invasive imaging techniques such as echocardiography, nuclear scintigraphy, computed tomography, and CMR .2D echocardiography is largely operator dependent and suffers from poor inter-study reproducibility.The complex geometry of the RV makes it difficult to accurately quantify remodelling before and after intervention. Nuclear scintigraphy and computed tomography (CT) are constrained by the need for ionizing radiation as well as the poor temporal resolution of the technique.Importantly, existing CMR analytics fail to exploit the full potential of the rich CMR image dataset, and do not yield information on regional RV remodelling, muscle stiffness and blood flow characterization.

Due to the challenges mentioned above, other than RV volumes and ejection fraction, other changes in RV shape and haemodynamics have yet to be considered in the official guidelines used to define eligibility for surgery and to quantify risk of operation. It is plausible that incorporation of additional variables that more comprehensively characterizes fine alterations in RV structure, function and haemodynamics in large risk-stratification models, such as the EuroSCORE and the Society of Thoracic Surgeons' Risk Calculator, may enhance risk stratification and prognostication.

Incorporating novel exploratory RV functional indices (e.g. curvedness, area strain) and computational methods (e.g. CFD, FSI simulations), and then correlating these with clinical and cardiopulmonary exercise test outcomes will allow investigators to have established an unprecedentedly sizeable and rich clinical imaging database that serves both as a touchstone for clinical reference, as well as a repository for future exploratory research.

Investigators tend to develop a comprehensive (BME) Research and Development platform for in-depth study of RV mechanics, blood flow and function in Congenital Heart Disease.

ELIGIBILITY:
Inclusion Criteria:

For patients with repaired tetralogy of Fallot

1. Survivors of TOF repair more than one year after repair
2. Aged: 12-80

For patients with pulmonary hypertension

1. Signed informed consent prior to initiation of any study mandated procedure
2. Age between 12 - 80 years
3. Patient with clinically suspected or known primary PH belonging to one of the following subgroups of the Updated Dana Point Clinical Classification Group 1 (at least 1 of the following a)Idiopathic (IPAH), or b)Heritable (HPAH), or c)Drug or toxin induced, or d)Associated (APAH) with one of the following: i.Connective tissue disease ii.Congenital heart disease

For Healthy volunteers

1. Aged :12-80
2. Asymptomatic and ambulant
3. Resting blood pressure <140/90 mmHg

Exclusion Criteria:

1. Non-cardiac illness with a life expectancy of less than 2 years
2. Previous heart, kidney, liver or lung transplantation
3. Contraindication to MRI examination

   1. Cardiac pacemaker
   2. Brain aneurysm or clips
   3. Electronic implants or prosthesis
   4. Eye metal foreign body injury
   5. Severe claustrophobia
   6. Severe renal impairment, glomerular filtration rate <30ml/min/1.73m2
4. Pregnancy

Additional exclusion criteria for healthy volunteers:

1. History of any major medical problems, any cardiovascular disease (such as hypertension or diabetes) or significant renal or lung disease (eg.COPD, Asthma, Pneumonia,Pulmonary embolism,Pulmonary edema,Respiratory tract infection,Bronchiolitis)
2. Concurrently taking any medications for cardiovascular disease (including hypertension)
3. Heavy smoking (over 5 sticks per day or who has quit smoking in less than 12 months and had smoked over 5 sticks per day)

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study will recruit 200 patients and 200 Healthy volunteers from across 3 sites at the following institutions:
  * National Heart Centre
  * National University Hospital
  * KK Women's and Children's Hospital
    200 Congenital Heart Disease Patients 200 Healthy Volunteer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Develop a comprehensive (BME) RnD platform for in-depth study of RV mechanics, blood flow and function in Congenital Heart Disease | 3 years
  This research will give an in-depth understanding of RV structure-function relationship, mechanics and haemodynamics. This is the foundation for rationale and physiologically-sound clinical decision-making in CHD monitoring and management. In addition, computational modelling of RV blood flow would be the best tool to optimize an individual solution to RV surgery and may ultimately improve surgical planning. This proposal is a pioneering study that can influence the research field and current management in preoperative, intraoperative, and post-operative interventions in CHD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Zhong Liang, Principal Investigator — Researcher
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - National Heart Centre, Singapore
  - KK Women's and Children's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Douglas PS, Pontone G, Hlatky MA, Patel MR, Norgaard BL, Byrne RA, Curzen N, Purcell I, Gutberlet M, Rioufol G, Hink U, Schuchlenz HW, Feuchtner G, Gilard M, Andreini D, Jensen JM, Hadamitzky M, Chiswell K, Cyr D, Wilk A, Wang F, Rogers C, De Bruyne B; PLATFORM Investigators. Clinical outcomes of fractional flow reserve by computed tomographic angiography-guided diagnostic strategies vs. usual care in patients with suspected coronary artery disease: the prospective longitudinal trial of FFR(CT): outcome and resource impacts study. Eur Heart J. 2015 Dec 14;36(47):3359-67. doi: 10.1093/eurheartj/ehv444. Epub 2015 Sep 1. PMID 26330417
- [Background] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Background] Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J, Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011 Nov 1;58(19):1989-97. doi: 10.1016/j.jacc.2011.06.066. PMID 22032711
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698
- [Background] Egidy Assenza G, Cassater D, Landzberg M, Geva T, Schreier J, Graham D, Volpe M, Barker N, Economy K, Valente AM. The effects of pregnancy on right ventricular remodeling in women with repaired tetralogy of Fallot. Int J Cardiol. 2013 Oct 3;168(3):1847-52. doi: 10.1016/j.ijcard.2012.12.071. Epub 2013 Jan 28. PMID 23369674
- [Background] Geva T, Sandweiss BM, Gauvreau K, Lock JE, Powell AJ. Factors associated with impaired clinical status in long-term survivors of tetralogy of Fallot repair evaluated by magnetic resonance imaging. J Am Coll Cardiol. 2004 Mar 17;43(6):1068-74. doi: 10.1016/j.jacc.2003.10.045. PMID 15028368
- [Background] Warnes CA. Adult congenital heart disease importance of the right ventricle. J Am Coll Cardiol. 2009 Nov 17;54(21):1903-10. doi: 10.1016/j.jacc.2009.06.048. PMID 19909869
- [Background] Kilner PJ, Geva T, Kaemmerer H, Trindade PT, Schwitter J, Webb GD. Recommendations for cardiovascular magnetic resonance in adults with congenital heart disease from the respective working groups of the European Society of Cardiology. Eur Heart J. 2010 Apr;31(7):794-805. doi: 10.1093/eurheartj/ehp586. Epub 2010 Jan 11. PMID 20067914
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Derived] Zhao X, Lee PT, Hu L, Tan RS, Chai P, Yeo TJ, Leng S, Ouyang R, Bryant JA, Teo LLS, van der Geest RJ, Yip JW, Tan JL, Zhong Y, Zhong L. Right Ventricular Restrictive Physiology Is Associated With Right Ventricular Direct Flow From 4D Flow CMR. JACC Asia. 2024 Oct 22;4(12):912-924. doi: 10.1016/j.jacasi.2024.08.019. eCollection 2024 Dec. PMID 39802994
- [Derived] Zhao X, Tan RS, Garg P, Chai P, Leng S, Bryant JA, Teo LLS, Yeo TJ, Fortier MV, Low TT, Ong CC, Zhang S, Van der Geest RJ, Allen JC, Tan TH, Yip JW, Tan JL, Hughes M, Plein S, Westenberg JJM, Zhong L. Age- and sex-specific reference values of biventricular flow components and kinetic energy by 4D flow cardiovascular magnetic resonance in healthy subjects. J Cardiovasc Magn Reson. 2023 Sep 18;25(1):50. doi: 10.1186/s12968-023-00960-x. PMID 37718441
- [Derived] Zhao X, Garg P, Assadi H, Tan RS, Chai P, Yeo TJ, Matthews G, Mehmood Z, Leng S, Bryant JA, Teo LLS, Ong CC, Yip JW, Tan JL, van der Geest RJ, Zhong L. Aortic flow is associated with aging and exercise capacity. Eur Heart J Open. 2023 Aug 26;3(4):oead079. doi: 10.1093/ehjopen/oead079. eCollection 2023 Jul. PMID 37635784
- [Derived] Zhao X, Leng S, Tan RS, Chai P, Yeo TJ, Bryant JA, Teo LLS, Fortier MV, Ruan W, Low TT, Ong CC, Zhang S, van der Geest RJ, Allen JC, Hughes M, Garg P, Tan TH, Yip JW, Tan JL, Zhong L. Right ventricular energetic biomarkers from 4D Flow CMR are associated with exertional capacity in pulmonary arterial hypertension. J Cardiovasc Magn Reson. 2022 Dec 1;24(1):61. doi: 10.1186/s12968-022-00896-8. PMID 36451198
- [Derived] Zhao X, Hu L, Leng S, Tan RS, Chai P, Bryant JA, Teo LLS, Fortier MV, Yeo TJ, Ouyang RZ, Allen JC, Hughes M, Garg P, Zhang S, van der Geest RJ, Yip JW, Tan TH, Tan JL, Zhong Y, Zhong L. Ventricular flow analysis and its association with exertional capacity in repaired tetralogy of Fallot: 4D flow cardiovascular magnetic resonance study. J Cardiovasc Magn Reson. 2022 Jan 3;24(1):4. doi: 10.1186/s12968-021-00832-2. PMID 34980199
- [Derived] Leng S, Tan RS, Guo J, Chai P, Zhang G, Teo L, Ruan W, Yeo TJ, Zhao X, Allen JC, Tan JL, Yip JW, Chen Y, Zhong L. Cardiovascular magnetic resonance-assessed fast global longitudinal strain parameters add diagnostic and prognostic insights in right ventricular volume and pressure loading disease conditions. J Cardiovasc Magn Reson. 2021 Apr 1;23(1):38. doi: 10.1186/s12968-021-00724-5. PMID 33789701
- See also: Clinical outcomes of fractional flow reserve. — https://www.ncbi.nlm.nih.gov/pubmed/26330417
- See also: Diagnostic accuracy of fractional flow reserve from anatomic CT angiography — https://www.ncbi.nlm.nih.gov/pubmed/22922562
- See also: Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. — https://www.ncbi.nlm.nih.gov/pubmed/22032711
- See also: Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). — https://www.ncbi.nlm.nih.gov/pubmed/22922698
- See also: The effects of pregnancy on right ventricular remodeling in women with repaired tetralogy of Fallot — https://www.ncbi.nlm.nih.gov/pubmed/?term=The+effects+of+pregnancy+on+right+ventricular+remodeling+in+women+with+repaired+tetralogy+of+fallot
- See also: Factors associated with impaired clinical status in long-term survivors of tetralogy of Fallot repair evaluated by magnetic resonance imaging — https://www.ncbi.nlm.nih.gov/pubmed/?term=Factors+associated+with+impaired+clinical+status+in+long-term+survivors+of+tetralogy+of+fallot+repair+evaluated+by+magnetic+resonance+imaging
- See also: Adult congenital heart disease importance of the right ventricle — https://www.ncbi.nlm.nih.gov/pubmed/?term=Adult+congenital+heart+disease+importance+of+the+right+ventricle.+J+Am+Coll+Cardiol+2009%3B
- See also: Recommendations for cardiovascular magnetic resonance in adults with congenital heart disease from the respective working groups of the European Society of Cardiology — https://www.ncbi.nlm.nih.gov/pubmed/?term=Recommendations+for+cardiovascular+magnetic+resonance+in+adults+with+congenital+heart+disease+from+the+respective+working+groups+of+the+European+Society+of+Cardiology
- See also: Computed tomography--an increasing source of radiation exposure — https://www.ncbi.nlm.nih.gov/pubmed/18046031